CLINICAL TRIAL: NCT05667194
Title: A Phase 1 Study to Assess the Safety ,Tolerability, Pharmacokinetics and Preliminary Antitumor Activity of KH617 After SAD and MAD Administration for Patients With Advanced Solid Tumors
Brief Title: Phase 1 Trial of KH617
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Honghe Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KH617
Record Dates: First submitted 2022-12-19; First posted 2022-12-28 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- KH617 dose 1 (Experimental): Three times (on days 1, 2, and 3) weekly for the first three consecutive weeks in a 28-day cycle
  Interventions: Drug: KH617
- KH617 dose 2 (Experimental): Three times (on days 1, 2, and 3) weekly for the first three consecutive weeks in a 28-day cycle
  Interventions: Drug: KH617
- KH617 dose 3 (Experimental): Three times (on days 1, 2, and 3) weekly for the first three consecutive weeks in a 28-day cycle
  Interventions: Drug: KH617
- KH617 dose 4 (Experimental): Three times (on days 1, 2, and 3) weekly for the first three consecutive weeks in a 28-day cycle
  Interventions: Drug: KH617
- KH617 dose 5 (Experimental): Three times (on days 1, 2, and 3) weekly for the first three consecutive weeks in a 28-day cycle
  Interventions: Drug: KH617

INTERVENTIONS:
Drug: KH617 — KH617 is s freeze-dried powder injection

SUMMARY:
KH617 is a injection used for advanced solid tumors which must be diluted with 5% Dextrose Injection.

ELIGIBILITY:
Inclusion Criteria:

* 1.Signed and dated written informed consent in accordance with International Council for Harmonisation - Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.

  2.Patient is male or female ≥18 years of age. 3.Patient must satisfy the following laboratory test results:

  a.Hemoglobin ≥9g/dL b.Platelet count ≥100×10^9/L c.Absolute neutrophil count≥1.5×10^9/L d.Albumin ≥3.0g/dL e.Total bilirubin ≤1.5×ULN f.Aspartate aminotransferase and alanine aminotransferase≤2.5×ULN g.Adequate renal function, defined as estimated serum creatinine clearance>50mL/minute calculated using the Cockcroft-Gault equation,urine protein<2+ or urine protein>2+ but 24-hour proteinuria<1g h.Prothrombin time, international normalized ratio, and activated partial thromboplastin time≤1.5×ULN (except for patients receiving anticoagulant therapy) 4.Patients who have fully recovered (defined as ≤grade 1 NCI-CTCAE 5.0) from all previous acute treatment-related toxic effects of previous cancer treatments prior to enrollment.

  5.Life expectancy at least 3 months. 6.Specific Inclusion Criteria
  1. Advanced Solid Tumors

     1. Patients with histopathology and/or cytology diagnosed as unresectable, locally advanced or metastatic malignant solid tumors for which there is no further standard treatment or for which the patient is not tolerated.
     2. Patient has at least one measurable or evaluable target lesion by RECIST 1.1.
     3. Patient has an ECOG status of 0 to 2.
  2. Brain Metastases

     1. Patient has at least one measurable or evaluable target lesion by RANO-BM.
  3. rGBM

     1. Patient with histopathology and/or cytology diagnosed advanced malignant adult diffuse glioma has unequivocal evidence of GBM recurrence/progression following completion of standard treatment.
     2. Patient has at measurable or evaluable target lesion by RANO.
     3. 4.Patient has a Karnofsky Performance score (KPS) ≥60.

        Exclusion Criteria:
* 1.Patient has received extensive radiation therapy. 2.Patients has the following infectious diseases:

  a.Hepatitis B surface antigen-positive and HBV-DNA test indicated active hepatitis B b.Active hepatitis c. C. AIDS or HIV antibody test is positive. d.Uncontrolled active infection. 3. Patient has a positive blood beta-HCG pregnancy test 7 days before the first administration (only for female with bearing potential ), or male and female with bearing potential who are unwilling to use adequate contraception for the duration of the study, and for a minimum of6 months after last dose of KH617.

  4. 11.Patient is currently pregnant or breastfeeding. 5. Patients with previous phrenoblabia history or currently phrenoblabia Including but not limited to schizophrenia, paranoia, phobias, obsessive-compulsive disorder, insomnia, Alzheimer's disease, behavioral volitional disorder, postpartum mental disorder, paranoid mental disorder, or organic psychosis.

  6. Patient has had another malignancy within the previous 5 years. 7. Patient has active cardiac or cerebrovascular disease. 8.Patient has participated in another investigational study using an investigational or marketed drug or device within 28 days.

  9. Patient has severe sensitivity/allergic reaction to KH617. 10.Patient has any other conditions that render them inappropriate for inclusion in the investigator's opinion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-12-26 (Actual); Primary Completion 2030-09 (Estimated); Study Completion 2031-08 (Estimated)

PRIMARY OUTCOMES:
MTD | 90 weeks
DLT | 90 weeks
RP2D | 154 weeks

SECONDARY OUTCOMES:
ORR | 154 weeks
PFS | 154 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Wenbin Li, Principal Investigator — Beijing Titan Hospital,Capital Medical University
Locations (1):
- Beijing Titan Hospital,Capital Medical University, Beijing, Beijing Municipality, China